CLINICAL TRIAL: NCT02354235
Title: Confirmatory Study of MT-2412 in Japanese Patients With Type 2 Diabetes (Add-on Study of Canagliflozin in Patients With Inadequate Glycemic Control on Teneligliptin)
Brief Title: Confirmatory Study of MT-2412 in Japanese Patients With Type 2 Diabetes (Add-on Study of Canagliflozin)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-2412-J03
Record Dates: First submitted 2015-01-29; First posted 2015-02-03 (Estimated); Results first posted 2018-08-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: MT-2412; MP-513; TA-7284; Teneligliptin; Canagliflozin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 3-(4-(4-(3-methyl-1-phenyl-1H-pyrazol-5-yl)piperazin-1-yl)pyrrolidin-2-ylcarbonyl)thiazolidine; Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canagliflozin + Teneligliptin (Experimental): Patients receive Canagliflozin for 24 weeks in combination with Teneligliptin.
  Interventions: Drug: Teneligliptin; Drug: Canagliflozin
- Placebo + Teneligliptin (Placebo Comparator): Patients receive placebo for 24 weeks in combination with Teneligliptin.
  Interventions: Drug: Teneligliptin; Drug: Placebo

INTERVENTIONS:
Drug: Teneligliptin
  Other Names: Tenelia, MP-513
Drug: Canagliflozin
  Other Names: Canaglu, TA-7284
  Arms: Canagliflozin + Teneligliptin
Drug: Placebo
  Arms: Placebo + Teneligliptin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of co-administration of Teneligliptin (MP-513) and Canagliflozin (TA-7284) once daily for 24 weeks in Japanese patients with Type 2 diabetes mellitus who are receiving treatment with Teneligliptin and have inadequate glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are 20 - 75 years old
* HbA1c of ≥7.0% and <10.5%
* FPG of ≤ 270 mg/dL
* Patients who are under dietary management and taking therapeutic exercise for diabetes over 8 weeks before run-in period

Exclusion Criteria:

* Patients with type I diabetes, diabetes mellitus resulting from pancreatic disorder, or secondary diabetes
* Patients with serious diabetic complications
* Patients with hereditary glucose-galactose malabsorption or primary renal glucosuria
* Patients with Class III/IV heart failure symptoms according to New York Heart Association (NYHA) functional classification
* Patients with severe hepatic disorder or severe renal disorder.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2015-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Kadowaki, MD, Study Director — Tokyo University; Kazuoki Kondo, MD, Study Director — Tanabe Pharma Corporation
Locations (3):
- Japan (3):
  - Reserch site, Kanto
  - Reserch site, Kinki
  - Reserch site, Tōhoku

REFERENCES:
- [Result] Kadowaki T, Inagaki N, Kondo K, Nishimura K, Kaneko G, Maruyama N, Nakanishi N, Iijima H, Watanabe Y, Gouda M. Efficacy and safety of canagliflozin as add-on therapy to teneligliptin in Japanese patients with type 2 diabetes mellitus: Results of a 24-week, randomized, double-blind, placebo-controlled trial. Diabetes Obes Metab. 2017 Jun;19(6):874-882. doi: 10.1111/dom.12898. Epub 2017 Mar 31. PMID 28177187

RESULTS

PARTICIPANT FLOW:
Groups:
- Canagliflozin+Teneligliptin: Canagliflozin for 24 weeks in combination with Teneligliptin
- Placebo+Teneligliptin: Placebo for 24 weeks in combination with Teneligliptin
Period: Overall Study
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Started | 70 | 68
Completed | 67 | 61
Not Completed | 3 | 7
Not completed — Adverse Event | 2 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Conflict with the stopping criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin | Total
Number analyzed (Participants) | 70 | 68 | 138
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 52 | 100
  >=65 years | 22 | 16 | 38
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 31
  Male | 54 | 53 | 107

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percentage of Glycated Hemoglobin (HbA1c)
Description: The change from baseline in percentage of HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at Week 24.
Time Frame: Baseline, 24 Weeks
Population: Full analysis set, last observation carried forward
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Number analyzed (Participants) | 70 | 68
percentage of HbA1c | -0.97 (0.10) | -0.10 (0.10)
Statistical Analysis 1: Comparison: Canagliflozin+Teneligliptin vs Placebo+Teneligliptin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -0.88, 95% CI 2-sided [-1.15 to -0.60], Standard Error of Mean 0.14

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Level
Description: The change from baseline in fasting plasma glucose level collected at Week 24.
Time Frame: Baseline, 24 Weeks
Population: Full analysis set, last observation carried forward. Outcome measure for one patient of each group was not assessed at a certain timepoint due to dropout.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Number analyzed (Participants) | 69 | 67
mg/dL | -34.9 (3.4) | 3.9 (3.5)
Statistical Analysis 1: Comparison: Canagliflozin+Teneligliptin vs Placebo+Teneligliptin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -38.8, 95% CI 2-sided [-48.5 to -29.2], Standard Error of Mean 4.9

3. Secondary Outcome: Percentage Change in Body Weight From Baseline
Description: The percentage change from baseline in body weight collected at Week 24.
Time Frame: Baseline, 24 Weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Number analyzed (Participants) | 69 | 67
percent change | -3.32 (0.31) | -0.99 (0.31)
Statistical Analysis 1: Comparison: Canagliflozin+Teneligliptin vs Placebo+Teneligliptin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -2.33, 95% CI 2-sided [-3.20 to -1.45], Standard Error of Mean 0.44

4. Secondary Outcome: Change From Baseline in the AUC(0-2h) for Postprandial Plasma Glucose (PPG)
Description: The change from Baseline in AUC(0-2h) for Postprandial Plasma Glucose collected at Week 24.
Time Frame: 0, 0.5, 1 and 2 hour postprandial, at Baseline and 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: hour*mg/dL
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Number analyzed (Participants) | 67 | 61
hour*mg/dL | -105.9 (7.6) | -5.6 (8.0)
Statistical Analysis 1: Comparison: Canagliflozin+Teneligliptin vs Placebo+Teneligliptin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -100.3, 95% CI 2-sided [-122.2 to -78.4], Standard Error of Mean 11.1

5. Secondary Outcome: Change From Baseline in 2-hour Postprandial Plasma Glucose Level
Description: The change from baseline in 2-hour postprandial plasma glucose level collected at Week 24.
Time Frame: 2 Hours Postprandial, at Baseline and 24 Weeks
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Number analyzed (Participants) | 67 | 61
mg/dL | -60.1 (4.9) | -9.2 (5.1)
Statistical Analysis 1: Comparison: Canagliflozin+Teneligliptin vs Placebo+Teneligliptin; Test type: Superiority; p < 0.001, ANCOVA; Least Squares Mean Difference = -50.9, 95% CI 2-sided [-64.9 to -36.9], Standard Error of Mean 7.1

ADVERSE EVENTS:
Arm/Group | Canagliflozin+Teneligliptin | Placebo+Teneligliptin
Serious Adverse Events (participants affected / at risk) | 1/70 | 2/68
Other Adverse Events (participants affected / at risk) | 13/70 | 11/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin+Teneligliptin (N=70) | Placebo+Teneligliptin (N=68)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Canagliflozin+Teneligliptin (N=70) | Placebo+Teneligliptin (N=68)
Nasopharyngitis (Infections and infestations) | 13 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other